CLINICAL TRIAL: NCT00006083
Title: A Phase III Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effects of Fragmin (5,000 IU Subcutaneously) in Preventing Catheter-Related Complications When Given Daily to Cancer Patients With Central Venous Catheters
Brief Title: Dalteparin to Prevent Complications in Cancer Patients Receiving Chemotherapy Through a Catheter
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Upjohn (Industry)
Responsible Party: John Glaspy, Jonsson Comprehensive Cancer center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CDR0000068075; UCLA-9910055; P-UPJOHN-98-FRAG-076; NCI-G00-1822
Record Dates: First submitted 2000-08-03; First posted 2004-05-26 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-07

CONDITIONS: Cervical Cancer; Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Precancerous/Nonmalignant Condition; Unspecified Adult Solid Tumor, Protocol Specific; Veno-occlusive Disease
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; monoclonal gammopathy of undetermined significance; recurrent adult Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage IB cervical cancer; Burkitt lymphoma; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; stage 0 chronic lymphocytic leukemia; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; unspecified adult solid tumor, protocol specific; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; chronic idiopathic myelofibrosis; essential thrombocythemia; untreated hairy cell leukemia; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; chronic myelomonocytic leukemia; T-cell large granular lymphocyte leukemia; acute undifferentiated leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; primary central nervous system lymphoma; prolymphocytic leukemia; primary systemic amyloidosis; veno-occlusive disease; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Precancerous Conditions; Hodgkin Disease; Monoclonal Gammopathy of Undetermined Significance; Lymphoma, T-Cell, Cutaneous; Burkitt Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Primary Myelofibrosis; Thrombocythemia, Essential; Leukemia, Hairy Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Leukemia, Myelomonocytic, Chronic; Leukemia, Large Granular Lymphocytic; Leukemia, Biphenotypic, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Immunoglobulin Light-chain Amyloidosis; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone | interventions — Dalteparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fragmin (Experimental): Fragmin at 5000 IU injected subcutaneously daily
  Interventions: Drug: Fragmin
- placebo (Placebo Comparator): placebo injected subcutaneously daily
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Fragmin — Fragmin at 5000 IU injected subcutaneously daily
  Arms: Fragmin
Other: placebo — placebo injected subcutaneously daily
  Arms: placebo

SUMMARY:
RATIONALE: The use of dalteparin may be able to prevent complications caused by the use of a catheter to supply chemotherapy to cancer patients. It is not yet known if dalteparin is effective in reducing these complications.

PURPOSE: Randomized phase III trial to determine the effectiveness of dalteparin in preventing catheter-related complications in cancer patients who are receiving chemotherapy through a catheter.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine if dalteparin will reduce the incidence of clinically significant catheter related complications (i.e., asymptomatic catheter related thrombosis) in cancer patients receiving chemotherapy through a central venous catheter.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to treatment center and catheter placement (proximal to axilla vs distal to axilla). Patients are randomized to one of two treatment arms. Arm I: Patients receive dalteparin subcutaneously (SC) daily. Arm II: Patients receive placebo SC daily. Treatment continues for 16 weeks or until catheter removal in the absence of unacceptable toxicity. Patients are followed for 30 days.

PROJECTED ACCRUAL: A total of 345 patients (230 in arm I and 115 in arm II) will be accrued for this study over 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy
* No more than 5 days since placement of central venous catheter for administration of chemotherapy
* Expected length of catheter use at least 16 weeks
* 18 and over
* Performance status: ECOG 0-2
* Life expectancy: At least 16 weeks
* Hematopoietic:
* Platelet count at least 100,000/mm3
* Absolute neutrophil count at least 1,500/mm3
* No known coagulopathy
* Hepatic: Bilirubin no greater than 2 times upper limit of normal (ULN) except in case of Gilbert's syndrome
* AST no greater than 3 times ULN (no greater than 5 times ULN in case of liver metastases)
* PT/PTT no greater than 1.5 times ULN Renal:
* Creatinine no greater than 2 times ULN Cardiovascular:
* HIV negative
* Must weigh at least 90 pounds
* At least 3 months since prior eye, ear, or CNS surgery Other:
* At least 30 days since prior aspirin, dipyridamole, unfractionated heparin, other low molecular weight heparins, or other anticoagulation therapy (except heparin flushing)

Exclusion Criteria:

* uncontrolled hypertension, unstable angina, or symptomatic congestive heart failure
* myocardial infarction in past 6 months
* uncontrolled cardiac arrhythmia Other:
* known hypersensitivity (including heparin induced thrombocytopenia) to dalteparin, heparin, or other low molecular weight heparins
* active uncontrolled infection, including existing catheter related infection
* CNS trauma in past 3 months
* retinal detachment in past 6 months
* mental incapacitation or psychiatric illness that would preclude study compliance
* other serious concurrent disease that would preclude study participation
* active gastrointestinal or genitourinary tract bleeding
* intracranial or intraocular hemorrhage in past year
* concurrent high dose chemotherapy with stem cell transplantation
* concurrent induction/consolidation chemotherapy for leukemia
* concurrent high dose chemotherapy with stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-04; Primary Completion 2000-11 (Actual); Study Completion 2000-11 (Actual)

PRIMARY OUTCOMES:
To determine if 5000 IU of Fragmin administered daily when compared to placebo will reduce the incidence of clinically relevant CRCs in cancer patients receiving chemotherapy by CVC | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John A. Glaspy, MD, MPH, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States